CLINICAL TRIAL: NCT01280357
Title: Study to Determine Substantial Equivalence of Electrohysterography (EHG) Monitoring to Tocodynanometer Monitoring
Brief Title: Accuracy and Reliability of Fetal Heart Rate and Uterine Contraction Monitoring Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Healthcare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MHL101801
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy; Habitual Aborter; Weeks of Gestation 37 or More
Keywords: Fetal Heart Rate (FHR); Uterine Activity (UA); Labor & Delivery
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitor Philips 50XM (K954351) (Active Comparator): CTG Fetal Monitor If not confident of Monica AN24 displayed data then remove Monica AN24 monitor and continue monitoring with Philips 50XM
  Interventions: Device: Philips 50XM
- Monica AN24 (K101801) (Experimental): EHG Fetal Monitor
  Interventions: Device: Monica AN24 (K101081)

INTERVENTIONS:
Device: Monica AN24 (K101081) — If not confident of Monica AN24 displayed data then remove Monica AN24 monitor and continue monitoring with Philips 50XM
  Other Names: Philips Series 50XM (K954351)
  Arms: Monica AN24 (K101801)
Device: Philips 50XM — If not confident of Monica AN24 displayed data then remove Monica AN24 monitor and continue monitoring with Philips 50XM
  Arms: Monitor Philips 50XM (K954351)

SUMMARY:
Clinical Investigation Protocol for a study designed to determine the equivalence of the Monica AN24 monitor to Philips 50XM for fetal heart rate (FHR) and uterine contraction (UC) monitoring during labor. The study will be carried out on subjects in the first and second stages of labor.

DETAILED DESCRIPTION:
The study is a prospective, randomized, single-center observational study designed to compare the Fetal Heart Rate (FHR) and Uterine Activity (UA) output data obtained by the Monica AN24 monitor during the first and second stages of labor to those generated by existing FDA-approved devices.Patients were enrolled at the facility but the patient details were removed from the results in order that the data could be randomized for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, age 15-40
* Term gestation (>36 completed weeks)
* Singleton fetus
* Active labor
* Vertex presentation
* Requiring internal monitoring

Exclusion Criteria:

* Clinical contraindication for Intra Uterine Pressure Catheter
* Major fetal malformation

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Cohen, MD, Study Director — Queens Hospital Centre
Locations (2):
- United States (2):
  - Queens Hospital Center, New York, New York
  - Temple University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was from Feb 2010 to Sept 2010 in a clinical setting at Queens Hospital Centre 82 - 68 164th Street Jamaica New York 11432
Pre-assignment Details: For all participants if there is any issue or exclusion from monitoring with the Monica AN24, fetal monitoring should continue using the Philips 50xm device
Groups:
- All Participants: during labor & delivery fetal heart rate, maternal heart rate and uterine contractions were monitored simultaneously by the Monia AN24 & the Philips 50XM
Period: Overall Study
Arm/Group | All Participants
Started | 60
Completed | 34
Not Completed | 26
Not completed — Excluded no internal monitoring | 14
Not completed — IInsufficient data/No data supplied | 12

BASELINE CHARACTERISTICS:
Groups:
- Monitor With the Philips 50XM, Remove Monica AN24: Intervention required if not confident of AN24 data is to remove the AN24 and continue monitoring with the predicate Tocco device
Arm/Group | Monitor With the Philips 50XM, Remove Monica AN24
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Secondary Outcome: The Mean Positive Percentage Agreement for Uterine Contractions Between the Monica AN24 & The Philips 50XM
Description: During labor and delivery uterine contractions were measured between the Monica AN24 & the philips 50XM, the waveforms of the two devices were measured to see the percentage of time they were in agreement
Time Frame: between 35 mins & 15hrs during first & second stage labor
Population: Of the remaining 34 participants in the clinical trials.The data was collected in the following manner.
  31 participants were used in FDA 6 way trial for Fetal Heart Rate (FHR) and Uterine Activity (UA) 2 participants were used in a 3 way trial for FHR
  1 participant was used in a 3 way trial for UA Equates to 33 files for FHR & 32 files for UA
Measure: Mean (95% Confidence Interval); unit: Positive Percentage Agreement (PPA)
Groups:
- All Participants: Continue monitoring with the Philips 50XM and disconnect the Monica AN24 monitor.
Arm/Group | All Participants
Number analyzed (Participants) | 32
Positive Percentage Agreement (PPA) | 96.61 [93.91 to 99.93]

2. Primary Outcome: The Mean Positive Percentage Agreement (PPA) for Fetal Heart Between Device 1 Monica AN24 & Device 2 Philips 50XM
Description: During Labor & delivery, fetal heart rate was measured between the Monica AN24 & the Philips 50XM and the waveforms of the 2 devices were measured to see the percentage of time they were in agreement.
Time Frame: during labor and delivery the waveforms were measured for between 35 minutes and 15 hours during the first and second stage of labour
Population: Of the remaining 34 participants in the clinical trials.The data was collected in the following manner.
  31 participants were used in a FDA 6 way trial for Fetal Heart Rate (FHR)and Uterine Activity (UA) 2 participants were uesd in a 3 way trial for FHR
  1 participant was used in a 3 way trial for UA Equates to 33 files for FHR & 32 files for UA
Measure: Mean (95% Confidence Interval); unit: Positive percantage agreement (PPA)
Groups:
- All Participants: all participants that had fetal heart rate measured with the Monica AN24 & the Philips 50XM
Arm/Group | All Participants
Number analyzed (Participants) | 33
Positive percantage agreement (PPA) | 84.85 [73.84 to 88.89]

3. Primary Outcome: The Mean Positive Percentage Agreement (PPA) for Maternal Heart Between Device 1 Monica AN24 & Device 2 Philips 50XM
Description: During Labor & delivery, maternal heart rate was measured between the Monica AN24 & the Philips 50XM and the waveforms of the 2 devices were measured to see the percentage of time they were in agreement.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Positive percantage agreement (PPA)
Groups:
- All Participants: all participants that had maternal heart rate measured with the Monica AN24 & the Philips 50XM
Arm/Group | All Participants
Number analyzed (Participants) | 33
Positive percantage agreement (PPA) | 99.3 [91.3 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored for the full length of the clinical trial, 6 months in total
Groups:
- Philips 50XM,; Monica AN24: Intervention required if not confident of AN24 data is to remove the AN24 and continue monitoring with the Philips 50XM
Arm/Group | Philips 50XM, | Monica AN24
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less